CLINICAL TRIAL: NCT06065683
Title: Acute Postoperative Pain Prevalence and Intensity in the First 72 Hours in Dessie Referral Hospital, Ethiopia: a Prospective Single-center Cohort Study
Brief Title: Acute Postoperative Pain Prevalence and Intensity in the First 72 Hours
Status: Completed | Type: Observational
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Sara Timerga, Lecturer, Wollo University
Other Study IDs: Acute pain
Record Dates: First submitted 2023-08-01; First posted 2023-10-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- T2 hour
  Interventions: Procedure: surgery
- T12 hour
  Interventions: Procedure: surgery
- T24 hour
  Interventions: Procedure: surgery
- T48 hour
  Interventions: Procedure: surgery
- T72 hour
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — Surgical procedures performed in the study period

SUMMARY:
Postoperative pain is poorly studied in developing countries. Severe pain after surgery remains a major problem, occurring in 50% to 70% of the patients. Differences exist across countries. Despite numerous published studies, the degree of pain following many types of surgery in everyday clinical practice is unknown. To improve postoperative pain treatment and develop procedure-specific, optimized pain-treatment protocols, the prevalence and severity of postoperative pain must first be identified.

This study aimed to determine the incidence and intensity of acute postoperative pain, to identify populations associated with a higher risk in order to guide resource allocation, and to investigate whether inexpensive analgesic modalities are currently utilized maximally.

DETAILED DESCRIPTION:
Postoperative pain management remains one of the major challenges in the care of surgical patients in many parts of the world. Despite improved care, studies show that postoperative pain continues to be inadequately treated and that patients still suffer moderate to severe pain after surgery. Despite an improved understanding of pain mechanisms, several risk factors, and advances in pain management strategies, postoperative pain continues to be a widespread and unresolved problem.

In Ethiopia, pain management is done in the traditional way, and pain control regimens vary from center to center and again from person to person in the same center due to a lack of pain management protocol. Overall pain management criteria used are not clear and sometimes decisions may be influenced by what is available in stock. Therefore, this research on the assessment of postoperative pain management provides information for clinicians to formulate protocols for the management of postoperative pain and for hospital managers in order to guide resource allocation to use limited resources efficiently and plan for optimum postoperative pain management.

In the study, the investigators used a numerical pain rating scale for pain immediately after surgery for the first 72 hours after surgery. The prevalence of mild, moderate, or severe pain and median pain scores were calculated. An evaluation will be performed at eight time points: at T2, T4, T8, T12, T24, T48, and T72. They consider 350 patients from all surgical wards. All surgical procedures were assigned to 5 well-defined groups. When a group contained less than 20 patients the data was excluded from the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Able to provide informed consent
* Able to verbalize or indicate pain by using a traditional verbal scale such as the numeric rating scale at the 2nd hr. of Post anesthesia care unit arrival.

Exclusion Criteria:

* Patients unable to self-report acute pain
* Patients with a history of chronic pain, moderate to high acute pain previous to surgery.
* Patients with a previous diagnosis of chronic cognitive impairment (Dementia, Alzheimer …)
* Patients with a previous diagnosis of Neurologic impairment (paraplegia, q quadriplegia…)
* The patients excluded from the study will be patients with mental and psychological problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients who will be undergo elective major abdominal, gynecologic, urologic, obstetric and orthopedic surgeries at Dessie comprehensive specialized hospital in the course of study period
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of postoperative pain in the first 72 hrs | 72 hours
  prevalence of postoperative pain , at 2nd, 4th, 8th, 12th, 24th, 48th and 72nd hr.

SECONDARY OUTCOMES:
Intensity of postoperative pain in the first 72 hrs. | 72 hours
  The intensity of postoperative pain in the first 72 hours assessed with numeric rating scale. NRS 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Timerga, Principal Investigator — Wollo University
Locations (1):
- Wollo Univeersity, Dessie, Ethiopia